CLINICAL TRIAL: NCT05617001
Title: Clinical Validation and Safety of the AC 12L ECG System Against a Standard of Care 12-Lead ECG (AC 12L ECG)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PRO-0012
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Kardia 12L — The purpose of this study is to collect clinical validation data to support an FDA submission for a 510(k) for the Kardia 12L hardware which enables the simultaneous diagnostic quality recording of all 6 limb leads and any chest lead. We will be recording both Leads V1 and V2 in a sequential fashion along with the V4 and Limb leads and a simultaneous 12-lead ECG to validate the hardware and a Deep Neural Network model which expands the 5 leads into a complete 12-lead ECG. The 12-lead ECG used for validation of the recordings and the 12-lead synthesis model is the GE Cardiosoft System which is FDA cleared.

SUMMARY:
AliveCor (www.alivecor.com) has developed an ECG device (KardiaMobile) that interfaces with iOS and Android smartphones and tablets. This ECG consists of a lightweight hardware case with two metal electrodes that can snap onto the back of the phone and a software application. By holding the right finger(s) on the right electrode and the left finger(s) on the left electrode, an electrical circuit is completed and a lead-I, 30 second rhythm strip is created. KardiaMobile and a newer device, KardiaMobile 6L, were approved by FDA for ECG rhythm recording. Recently, AliveCor developed a new device: Kardia 12L to record 12-lead ECGs. However, the data generated from the new device has not yet been validated for accuracy. The specific aim of this study is to evaluate the accuracy and safety of the AC 12L ECG System. The ECGs collected by the AC 12L ECG System will be compared to simultaneous standard- of-care 12-lead ECG, recorded using the GE CardioSoft 12-lead ECG System. The ECGs will be analyzed for accuracy based on statistical difference using root-mean-square error, and cross correlation between the simultaneous 10 second recordings as well as the median beats of all 12 leads.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 years or older
* Ability to remain supine for a conventional 12 lead AliveCor 12L ECG recording for approximately 15 minutes

Exclusion Criteria:

* Open chest wounds or recent (<30 days) surgery to the chest or abdomen
* Absence of any limb that would require modification of the lead set-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-10-04 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Agreement on QRS width between Kardia 12L and ECG | 30 seconds
  Quantitative analysis on QRS width will be performed on the median-beat ECGs derived from the recorded ECGs from the device as well as 12-lead ECG for each study participant
Agreement on PR interval between Kardia 12L and ECG | 30 seconds
  Quantitative analysis on PR interval will be performed on the median-beat ECGs derived from the recorded ECGs from the device as well as 12-lead ECG for each study participant
Agreement on AT interval between Kardia 12L and ECG | 30 seconds
  Quantitative analysis on AT interval will be performed on the median-beat ECGs derived from the recorded ECGs from the device as well as 12-lead ECG for each study participant

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Stavrakis, MD, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided